CLINICAL TRIAL: NCT06424379
Title: Study of Clinical, Histological, Immunohistochemical and Molecular Impact of BCL6 Gene Rearrangement in Most Prevalent Non-Hodgkin Lymphomas
Brief Title: BCL6-rearrangements Implications in Non-Hodgkin Lymphomas.
Acronym: BCL6-RINHL
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0515
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Non Hodgkin Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Diffuse Large B Cell Lymphoma
Keywords: Non Hodgkin Lymphoma; BCL6 gene rearrangement; Next generation sequencing
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The samples analyzed will have been collected as part of routine medical care for each patient before inclusion in the study.
  These are formalin-fixed, paraffin-embedded (FFPE) tissue samples. They will be packaged and stored in the Biological Resources Center of the Hospices Civils de Lyon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Follicular lymphomas with BCL6 gene rearrangement: Diagnoses of follicular lymphomas based on the last World Health Organization (WHO) classification of haematolymphoid tumours at the time of occurrence of the disease. Fluorescence in situ hybridization (FISH) utilizes Vysis' Dual-Color Break-Apart Rearrangement Probes to detect BCL6 gene alterations. FISH patterns have been interpreted following established protocols.
  Interventions: Other: Histopathological analysis; Genetic: Molecular analysis
- Marginal zone lymphomas with BCL6 gene rearrangement: Diagnoses of marginal zone lymphomas based on the last WHO classification of haematolymphoid tumours at the time of occurrence of the disease. FISH utilizes Vysis' Dual-Color Break-Apart Rearrangement Probes to detect BCL6 gene alterations. FISH patterns have been interpreted following established protocols.
  Interventions: Other: Histopathological analysis; Genetic: Molecular analysis
- Diffuse large B-cells lymphomas with BCL6 gene rearrangement: Diagnoses of diffuse large B-cells lymphomas based on the last WHO classification of haematolymphoid tumours at the time of occurrence of the disease. FISH utilizes Vysis' Dual-Color Break-Apart Rearrangement Probes to detect BCL6 gene alterations. FISH patterns have been interpreted following established protocols.
  Interventions: Other: Histopathological analysis; Genetic: Molecular analysis

INTERVENTIONS:
Other: Histopathological analysis — Morphological analysis will include the description of architectural patterns and cytological features on formalin-fixed and paraffin-embedded (FFPE) tissue samples retrieved from the routine diagnostic archives of the Pathology Department of the University Hospital Lyon Sud.
  A panel of immunohistochemical staining will be analyzed including CD20, CD3, CD10, Bcl-6, Bcl-2, CD5, CD23, CD38, MUM1, Ig kappa, Ig lambda, MEF2B, LMO2, MNDA, IRTA1, P53, CMYC and Ki67 . /MIB1. Diffuse large B-cells lymphomas will be classified into two distinct subgroups: centro-germinative (GC) and non-centro-germinative (nGC), using the Hans algorithm.
Genetic: Molecular analysis — Next-generation sequencing (NGS) analysis will be performed on FFPE tissue samples retrieved from the routine diagnostic archives of the Pathology Department of the University Hospital Lyon Sud. A panel of 73 genes dedicated to lymphoma diagnosis determined by a consensus of French Lysa experts will be used. The identification of genetic variants will be followed by the attribution of pathogenicity class in accordance with the guidelines for validation of NGS-based oncology panels.
  RNA extraction will classify DLBCLs into two distinct subgroups: germinal-centre B-cell-like (GCB-DLBCL) and activated B-cell-like (ABC-DLBCL).

SUMMARY:
Non-Hodgkin lymphomas (NHLs) constitute a heterogeneous group of malignant neoplasms, with diverse clinical behaviors and distinct pathologic and molecular characteristics. Among these lymphomas, follicular lymphomas (FLs), marginal zone lymphomas (MZLs) and diffuse large B-cell lymphomas (DLBCLs) emerge as the most prevalent entities. While FL and MZL are representative of indolent B-cell lymphomas, characterized by a slow progression of the disease and favorable clinical outcomes, DLBCL stands out as an aggressive lymphoma, often occuring from the transformation of a pre-existing indolent lymphoma.

Chromosome translocations are a hallmark of some NHL subtypes, offering insights into their molecular pathogenesis. For instance, the conventional FL is genetically characterized by the t(14;18) chromosomal translocation, found in 85-90% of cases, resulting in sustained elevation of the antiapoptotic protein B-cell lymphoma 2 (BCL2). However, certain FL cases lack BCL2 translocations and exhibit distinct clinical, morphological and phenotypical features with genetic heterogeneity.

A subset of BCL2-negative FLs displays rearrangements within chromosomal region 3q27, inducing abnormal modulation of B-cell lymphoma 6 (BCL6) expression. The BCL6 gene plays a critical role in germinal center development and B-cell differentiation. Previous investigations indicate that BCL6 rearrangements (BCL6-R) manifest distinct pathological and genetic features, diverging from classical FL presentations.

FLs carrying BCL6-R commonly share a specific CD10- Bcl-2- Bcl-6+ phenotype, often accompanied by a monocytoid component and increased frequency of diffuse architectural patterns. Patients with BCL6-R tend to exhibit advanced clinical stages and complex genetic profiles.

MZLs present differential diagnostic challenges due to shared monocytoid components, phenotypes traits, and common genetic features. The similarities observed between BCL6-R FL and MZL suggest a convergence in both morphological and genetic aspects, leading to intricate differentiation. Traditionally, these indolent NHLs with BCL6-R were categorized as FL and incorporated into the FL category in the WHO classification. However, few studies highlight the occurrence of BCL6-R in MZLs. This observation gives rise to the hypothesis that indolent NHLs exhibiting BCL6-R might correspond to a continuum comprising both FL and MZL.

Additionally, BCL6-R has been frequently documented in DLBCL cases with residual MZL component. These DLBCL cases might display a mutational profile reminiscent of MZL. This suggests a plausible origin of BCL6-R DLBCL from indolent BCL6-R MZLs or BCL6-R FLs cases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of non-Hodgkin's lymphoma at anatomy and cytology department of Lyon Sud hospital
* Rearrangement of the BCL6 gene detected by FISH analysis
* Diagnostic of the disease between january 2016 and december 2023

Exclusion Criteria:

* Patients diagnosed with primary cutaneous centrofollicular B lymphoma, composite lymphoma, anaplastic B lymphoma or primary B lymphoma of the mediastinum.
* Presence of a rearrangement of the BLC2 gene or the CMYC gene in FISH
* Presence of a non-significant BCL6 gene rearrangement (<5% of rearranged cells)

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with non-Hodgkin lymphoma from the routine diagnostic archives of the pathology department of CHU Lyon Sud between January 2016 and August 2023 and with BCL6-R detected by FISH analysis will be included in the study. A cohort of 135 cases will be assembled and subjected to the analysis.
  This dataset will be reviewed by two haematopathologists to ensure the inclusion of the most relevant cases. Selection will favor cases with substantial histological material and available clinical, immunophenotypic and cytogenetic data. Comparative assessments will be conducted between distinct subtypes of NHL exhibiting BCL6-R, including FLs, MZLs, and DLBCLs.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of LF and MZL with BCL6-R. | The primary outcome will be analyzed retrospectively, or through study completion, an average of 1 year
  An examination of morphological attributes, including tissue architecture and cellular patterns will be performed on LF and MZL with BCL6-R. An extended immunohistochemical staining panel employing incorporated novel centro-germinative markers (LMO2 and MEF2B) and recently identified MZL-specific markers (IRTA1 and MNDA) is planned.
Comparison of LF and MZL with BCL6-R. | The primary outcome will be analyzed retrospectively, or through study completion, an average of 1 year
  Fluorescence in situ hybridization (FISH) will be employed for cytogenetic evaluation to detect BCL2 and BCL6 gene rearrangements. In parallel, targeted next-generation sequencing (NGS) analysis will enable genetic variant detection.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Lyon Sud - HCL, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No